CLINICAL TRIAL: NCT00628524
Title: Prospective Investigation of the Influence of Triglyceride Tolerance on Cardiovascular Outcomes in Patients With Coronary Artery Disease
Brief Title: Homburg Cream & Sugar Study
Acronym: HCS
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: HCS Study
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2013-12

CONDITIONS: Coronary Artery Disease; Diabetes; Metabolic Syndrome; Glucose Tolerance; Hyperlipidemia
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus; Metabolic Syndrome; Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: > 500 consecutive patients with coronary artery disease fulfilling eligibility criteria.

SUMMARY:
The purpose of this study is to prospectivly analyze the correlation of triglyceride tolerance and glucose tolerance with cardiovascular morbidity and mortality in patients with stable coronary artery disease within 18 months and to determine, whether measurement of triglyceride tolerance can discriminate patients at risk for cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Stable CAD

Exclusion Criteria:

* Acute Coronary Syndrom
* Relevant Arrhythmias
* Severe valvular heart disease
* Decompensated heart failure
* Severe inflammtory disease (infectious, rheumatoid)
* Metabolic diseases (e.g. thyroid)
* Inability to swallow
* Liver or kidney failure
* Lactose intolerance
* Fat intolerance (e.g. chronic pancreatitis, gall stones)
* Malignant Disease
* Psychiatric Diseases (including alcohol / drug abuse)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: > 500 consecutive patients with stable coronary artery disease being treated in the cardiology department of the university hospital.
Sampling Method: Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2008-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Parameters of triglyceride tolerance and glucose tolerance in correlation to cardiovascular events, cardiovascular mortality, total mortality. | 48 months after inclusion.

SECONDARY OUTCOMES:
Waist-to-Hip ratio, nutrition protocol, physical activity, non-invasive endothelial function, body fat composition, other biomarkers of lipid and glucose metabolism. | Directly after inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Laufs, MD, Principal Investigator — University Hospital, Saarland
Locations (1):
- University Hospital Homburg / Saar - Cardiology Department, Homburg, Saarland, Germany

REFERENCES:
- [Result] Werner C, Filmer A, Fritsch M, Groenewold S, Graber S, Bohm M, Laufs U. Risk prediction with triglycerides in patients with stable coronary disease on statin treatment. Clin Res Cardiol. 2014 Dec;103(12):984-97. doi: 10.1007/s00392-014-0740-0. Epub 2014 Jul 11. PMID 25012240
- [Derived] Katzmann JL, Werner CM, Stojakovic T, Marz W, Scharnagl H, Laufs U. Apolipoprotein CIII predicts cardiovascular events in patients with coronary artery disease: a prospective observational study. Lipids Health Dis. 2020 May 30;19(1):116. doi: 10.1186/s12944-020-01293-9. PMID 32473635
- [Derived] Hoffmann MM, Werner C, Bohm M, Laufs U, Winkler K. Association of secreted frizzled-related protein 4 (SFRP4) with type 2 diabetes in patients with stable coronary artery disease. Cardiovasc Diabetol. 2014 Nov 19;13:155. doi: 10.1186/s12933-014-0155-2. PMID 25408147